CLINICAL TRIAL: NCT00735215
Title: Faslodex Registry: a Belgian Observational Study to Evaluate the Use of Fulvestrant in Current Clinical Practice
Brief Title: Faslodex Registry: Fulvestrant in Current Clinical Practice
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Anna Chioti, MD, Therapeutic Area Leader Oncology, AstraZeneca Belgium
Other Study IDs: NIS-OBE-FAS-2008/1
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast cancer,; fulvestrant,; postmenopausal,; women; locally advanced,; hormone receptor-positive.
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The sequential administration of endocrine therapies to patients with advanced breast cancer requires the availability of therapies with different modes of actions, so that tumours developing resistance to one agent are not cross resistant to another. Because of its mechanism of action, fulvestrant is distinct from other hormonal therapies, which therefore limits the possibility of cross-resistance with other therapies such as tamoxifen and the aromatase inhibitors (AIs)

* In this way, patients may benefit from an extended period of endocrine treatment, which has considerable tolerability and quality-of-life advantages over cytotoxic chemotherapy.
* In Belgium, fulvestrant is indicated for treating postmenopausal women with hormone receptor-positive locally advanced or metastatic breast cancer with recurrence during or after adjuvant anti-oestrogen therapy or disease progression during anti-oestrogen treatment. However, little information is currently available on how fulvestrant is actually being used by physicians in Belgium. The optimum sequence of endocrine treatment for advanced breast cancer has yet to be defined and may depend on certain patient or disease characteristics.

Fulvestrant has been granted reimbursement by the Belgian Health authorities (RIZIV/INAMI) with the recommendation to collect the real life data necessary to assess the patients' breast cancer treatment history that may influence the actual endocrine treatment sequence according to physicians current clinical practice..

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with hormone receptor-positive locally advanced or metastatic breast cancer

Exclusion Criteria:

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Woman with post-menopausal breast cancer.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-10; Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
to collect real life data on the use of fulvestrant in clinical practice in Belgium. Previous therapies (hormonal and chemo) for breast cancer and for advanced breast cancer will be documented for each patient. | Visit 1, Visit 2

SECONDARY OUTCOMES:
Document treatment during observation period and number of fulvestrant injections | Visit 1, Visit 2
Document reasons for fulvestrant treatment discontinuation | Visit 2

CONTACTS AND LOCATIONS:
Overall Officials: Neven P Prof, Study Director — KUL
Locations (12):
- Belgium (12):
  - Research Site, Antwerp
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Kortrijk
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Namur
  - Research Site, Ostend
  - Research Site, Roeselare
  - Research Site, Turnhout
  - Research Site, Wilrijk